CLINICAL TRIAL: NCT02670720
Title: OPuS-4: An Open-label Study to Evaluate the Long-term Safety of Avoralstat in Subjects With Hereditary Angioedema
Brief Title: Open-label, Long-term Safety Study of Avoralstat in Subjects With Hereditary Angioedema
Acronym: OPuS-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: preceding efficacy study of avoralstat in its current formulation was not significant and does not support continued development
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCX4161-303
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Hereditary Angioedema; HAE
Keywords: BCX4161; avoralstat; HAE; hereditary angioedema; prophylaxis
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — avoralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- avoralstat (Experimental): Five avoralstat capsules (100 mg) to be taken three times daily by mouth
  Interventions: Drug: avoralstat

INTERVENTIONS:
Drug: avoralstat
  Other Names: BCX4161

SUMMARY:
This is an open-label study designed to evaluate the long-term safety of prophylactic avoralstat (500 mg three times daily) when given to approximately 150 patients with hereditary angioedema (HAE) for a duration of up to 72 weeks. The study will also evaluate the long-term efficacy and impact on quality of life of avoralstat prophylactic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females age ≥ 18 years.
* Provide written, informed consent.
* Prior completion of an avoralstat therapeutic study OR a confirmed diagnosis of HAE Type 1 or HAE Type 2.
* Access to appropriate medication for the treatment of acute HAE attacks.
* Adequate contraception.

Exclusion Criteria:

* Females who are pregnant or breast feeding.
* Clinically significant medical condition or medical history.
* Abnormal screening ECG, laboratory or urinalysis finding that is clinically significant.
* Investigational drug exposure within 30 days (except avoralstat).
* History of or current alcohol or drug abuse.
* HIV or active HBV or HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who discontinue due to a treatment-emergent adverse event, who experience a treatment-emergent serious AE, who experience a Grade 3 or 4 AE and who experience Grade 3 or 4 laboratory abnormalities | Up to 72 weeks

SECONDARY OUTCOMES:
Angioedema attack rate (subject-reported HAE attacks normalized for time on study) | Up to 72 weeks
Durability in response (assessed as subject-reported HAE attacks) | change over time through 72 weeks
Proportion of subjects who discontinue avoralstat with a reason of lack of efficacy | Up to 72 weeks
Quality of life as determined by the EQ-5D-5L | Up to 72 weeks
Quality of life as determined by the Angioedema Quality of Life Questionnaire | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Farkas, MD, PhD, DSc, Principal Investigator — Semmelweis University
Locations (3):
- Leuven, Belgium
- France (2):
  - Grenoble
  - Lille